CLINICAL TRIAL: NCT05139446
Title: Reproductive Outcomes Following Uterine Septum Resection- a Bicentric Retrospective Study
Brief Title: Reproductive Outcomes Following Uterine Septum Resection
Acronym: UTER-SEPTUM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8070
Record Dates: First submitted 2021-10-13; First posted 2021-12-01 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2021-10

CONDITIONS: Uterine Septum
Keywords: uterine septum; Hysteroscopic septum resection; Metroplasty; Subfertility; Infertility; Preterm delivery; Spontaneous abortion
MeSH Terms: conditions — Septate Uterus; Infertility; Premature Birth; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, there is little data to validate the performance of surgical hysteroscopies in the case of septate uterus, particularly in the case of incidental discoveries. Clinical practice and the experience of teams leads to propose this procedure, but strong evidence for this recommendation is lacking and there is an urgent need for solid data.

A recent randomized trial contradicts this recommendation, but the methodology is questionable on several points.

Investigators wished to associate 2 reference centers with current practice and expertise on this procedure in order to have a cohort of many patients and to have more powerful results.) Investigators purpose a retrospective observational data-based study. The aim is to describe the profile of patients with a partitioned uterus in terms of obstetrical history and to study the consequences of uterine partition resection in terms of obstetrical prognosis (live births, at term, number of miscarriages or premature births).

The aim of this study is to take into account the evaluation of the surgical hysteroscopy gesture by postoperative imaging with in particular the indication of a resection in several stages in case of residual postoperative septum.

ELIGIBILITY:
Inclusion criteria:

Major female (≥18 years old) To be an operating patient at the strabourg university hospital or Bicetre Hospital between January 2009 and December 2019.

Exclusion criteria:

Particular clinical forms of the disease, (associated enlargement metroplasties, other uterine maformations) Minor patients, patients under guardianship

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Major female (≥18 years old) being an operating patient at the strabourg university hospital or Bicetre Hospital between January 2009 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Retrospective study of the uterine septum resection technique by operative hysteroscopy | Files analysed retrospectively from January 01, 2009 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France